CLINICAL TRIAL: NCT01947972
Title: Individualized Maternal Milk Fortification for Feeding the Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Elisavet Parlapani, Dietitian - phD candidate, Aristotle University Of Thessaloniki
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IKY5721
Record Dates: First submitted 2013-09-10; First posted 2013-09-23 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Metabolic Syndrome
Keywords: preterm neonate; tailored fortification; nutrition; maternal breast milk composition
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- protein intake of 4g/kg/d (Other): Tailored protein fortification and nutritional status of preterm neonate. 4.5g protein per kg for preterms with body weight less than 1000g and 4g protein per kg for preterms with body weight more than 1000g, after human milk analysis. Intervention regards protein supplementation to fulfil the exact protein needs of preterms
  Interventions: Dietary Supplement: Tailored protein fortification

INTERVENTIONS:
Dietary Supplement: Tailored protein fortification — 4-4.5g of protein/kg/d

SUMMARY:
Neonatal nutrition has to face a contradictory and conflicting nutritional regimen like a high percentage of amino acids from the first day of life in order to achieve normal neurodevelopment versus metabolic complications (insulin resistance, hyperglycemia, increased visceral fat) that this type feeding, in conjunction with complexity of prematurity, is likely to cause. Current study aims to investigate is whether individualized fortification of breast milk protein, based on the mother's milk protein content and targeting the recommended daily protein requirements, is associated with better nutrition, growth, biochemical and endocrine markers associated with the nutrition of preterm low birth weight neonates, compared to the standard fortification of human milk.

DETAILED DESCRIPTION:
Proteins are of the most important macromolecules in living organisms participating in almost all biological processes. Premature infants are forced to adapt to a new (extrauterine) environment where supply of nutrients, including amino acids, from mother ceases abruptly. Consequently, the aim of neonatologist is the appropriate, quantitatively and qualitatively nutritional support, to promote brain development, achieve normal endocrine and metabolic function, maintain a growth rate similar to the intrauterine one avoiding extrauterine growth restriction during postnatal period and at the same time encouraging the analogue modulation of body composition (increased muscle mass, decrease body fat, hydration).

Malnutrition or inadequate nutrition of preterm infant which remains undiagnosed and without proper treatment could have serious consequences on psychomotor development and metabolic activity. Indeed, 75% of low birth weight premature infants exhibit extrauterine growth restriction at discharge, even when they have achieved growth equal to the considered satisfactory, ie 15g/kg/day.

Beyond anthropometrics differences between preterm and full-term newborns, body composition varies as well. Preterms have higher percentage of body fat and decreased muscle mass at term time compared with full term neonates. However, it has not been clarified whether this differentiation is harmful predisposing to chronic diseases later in childhood or adult life (eg. obesity, metabolic syndrome).

ELIGIBILITY:
Inclusion Criteria:

* Infants with gestational age ≤ 34weeks
* very low birth weight (≤ 1500g)

Exclusion Criteria:

* maternal health problems contradicting breastfeeding
* genetic or chromosomal abnormalities
* metabolic contraindications for increased amount of protein

Ages: 24 Hours to 5 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2013-10; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Mean protein intake per kg of body weight between the groups | participants will be followed until discharge and at 40 weeks post gestational age

SECONDARY OUTCOMES:
growth assessment differences between groups | participants will be followed until discharge and at 40 weeks post gestational age
  Anthropometric differences in body length, head circumference, body weight gain/kg, mid arm circumference
Differences in bioelectrical impedance between groups | participants will be followed until discharge and at 40 weeks post gestational age
Mean daily dietary intake of mothers and correlation with macronutrients of their's breast milk | from the moment of intervention, at least once in 10days, and until the end of intervention
Biochemical (lipidemic profile differences) between groups | at 36weeks post conceptual age and follow-up at 40 weeks postconceptual age

CONTACTS AND LOCATIONS:
Overall Officials: Elisavet Diamanti, Dr, Principal Investigator — AUTH
Locations (1):
- Hippokration Hospital Thessaloniki, Thessaloniki, Greece